CLINICAL TRIAL: NCT05809440
Title: The Effectiveness of Single Session 20-minute Mindful Breathing in Symptom Control in Kidney Transplant Recipients: a Randomised Controlled Trial
Brief Title: Effectiveness of 20m-MB in KTR Symptom Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, A/Prof. Dr. Ng Kok Peng, Consultant Nephrologist, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020116-9206
Record Dates: First submitted 2022-09-25; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Transplant;Failure,Kidney
Keywords: transplant; mindfulness; mindful breathing

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, non-blinded, randomized controlled trial conducted at the University of Malaya Medical Centre, Malaysia. Patients were recruited from the transplant clinic, the renal day care unit and the nephrology ward. Participants were randomly assigned to either intervention or control based on computer generated random number with 1:1 allocation ratio. Allocations were concealed with sealed envelopes.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A 20-minute mindful breathing session guided by a trained medical doctor. The session consisted of four 5-minute breathing exercises done consecutively. Participants were instructed to close their eyes and bring their attention to their breathing, and re-direct their attention back to their breathing once they were distracted.
  Interventions: Other: 20-minute mindful breathing session
- Control Group (No Intervention): No intervention was provided for control group.

INTERVENTIONS:
Other: 20-minute mindful breathing session — A 20-minute mindful breathing session guided by a trained medical doctor. The session consisted of four 5-minute breathing exercises done consecutively. Participants were instructed to close their eyes and bring their attention to their breathing, and re-direct their attention back to their breathing once they were distracted.
  Arms: Intervention Group

SUMMARY:
To study the effectiveness of single session 20-minute mindful breathing in symptom control in kidney transplant recipients.

DETAILED DESCRIPTION:
Patients undergoing kidney transplant follow ups in our center are screened based on recruitment criteria. Patients who fulfilled the incusion criteria are recruited. Intervention involves a 20-minute mindful breathing session with uniform script performed by trained personal, while control arm involves standard care without intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult renal transplant patients aged 18 years and older
* At least one symptom scoring ≥ 4/10 based on the Edmonton Symptom Assessment Scale (ESAS)

Exclusion Criteria:

* Dialysis-dependent
* Medically unstable
* Having serious pre-existing mental health issues

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Participant-rated Edmonton Symptom Assessment Scale (ESAS) scores at 0 minute and 20 minute | 20 minutes
  ESAS is a validated scale to assess 10 symptoms commonly experienced by patients, which are: pain, fatigue, nausea, depression, anxiety, drowsiness, shortness of breath, anorexia, other symptoms, and feelings of well-being. The severity of each symptom was rated on a numerical scale of 0 to 10 (0 = no symptom; 10 = worst possible symptom).

SECONDARY OUTCOMES:
Within-group comparison of Edmonton Symptom Assessment Scale (ESAS) scores at 0 minute and 20 minute | 20 minutes
  Statistical anaylsis done using paired t-tests.
Between-group comparison of changes in Edmonton Symptom Assessment Scale (ESAS) scores | 20 minutes
  Statistical anaylsis done using independent sample t-tests

CONTACTS AND LOCATIONS:
Overall Officials: Seng Beng Tan, MBBS, Principal Investigator — University of Malaya; Kok Peng Ng, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not shared.

REFERENCES:
- [Result] Afshar M, Rebollo-Mesa I, Murphy E, Murtagh FE, Mamode N. Symptom burden and associated factors in renal transplant patients in the U.K. J Pain Symptom Manage. 2012 Aug;44(2):229-38. doi: 10.1016/j.jpainsymman.2011.08.005. Epub 2012 May 10. PMID 22578312
- [Result] Yong DS, Kwok AO, Wong DM, Suen MH, Chen WT, Tse DM. Symptom burden and quality of life in end-stage renal disease: a study of 179 patients on dialysis and palliative care. Palliat Med. 2009 Mar;23(2):111-9. doi: 10.1177/0269216308101099. Epub 2009 Jan 19. PMID 19153131
- [Result] Taylor K, Chu NM, Chen X, Shi Z, Rosello E, Kunwar S, Butz P, Norman SP, Crews DC, Greenberg KI, Mathur A, Segev DL, Shafi T, McAdams-DeMarco MA. Kidney Disease Symptoms before and after Kidney Transplantation. Clin J Am Soc Nephrol. 2021 Jul;16(7):1083-1093. doi: 10.2215/CJN.19031220. Epub 2021 Jun 18. PMID 34597266
- [Result] Wang H, Du C, Liu H, Zhang S, Wu S, Fu Y, Zhao J. Exploration of symptom experience in kidney transplant recipients based on symptoms experience model. Qual Life Res. 2020 May;29(5):1281-1290. doi: 10.1007/s11136-019-02404-5. Epub 2020 Jan 2. PMID 31898113

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/40/NCT05809440/Prot_SAP_000.pdf